CLINICAL TRIAL: NCT00167518
Title: Phase II/III Intravitreal Triamcinolone for Treatment of Clinically Significant Diabetic Macular Oedema That Persists After Laser Treatment
Brief Title: Intravitreal Triamcinolone for Clinically Significant Diabetic Macular Oedema That Persists After Laser Treatment (TDMO)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JDRF 1-2003-767; ORIA Esme Anderson Grant; Sydney Eye Hospital Foundation
Record Dates: First submitted 2005-09-05; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-01

CONDITIONS: Diabetic Macular Oedema
Keywords: Diabetic macular oedema; Triamcinolone acetate; Intravitreal injection; Clinical trial; Laser treatment
MeSH Terms: interventions — Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone acetate

SUMMARY:
The trial will test the hypothesis that an intravitreal injection of triamcinolone is safe and efficacious for patients with clinically significant diabetic macular oedema that is recalcitrant to conventional laser therapy

DETAILED DESCRIPTION:
Diabetic retinopathy is a common cause of severe loss of visual and the most common cause of legal blindness in individuals between the ages of 20 and 65 years in developed countries. Swelling of the central retina, or "macular oedema" is the commonest cause of visual loss in diabetic retinopathy.

Diabetic macular oedema is treated with laser coagulation to the macular area according to established guidelines which take into account the extent of the leak and its proximity to the centre of the macula, the "fovea". This treatment does not, however, always work and is inherently destructive.

Intravitreal injection of crystalline steroids has been proposed as a new modality to treat clinically significant diabetic macular oedema.

To determine by means of a prospective, double-masked, randomised, placebo-controlled trial to determine whether an intravitreal injection of triamcinolone three months or more after focal or grid laser photocoagulation for clinically significant diabetic macular oedema will improve the visual acuity of eligible eyes. OCT will be used in addition to visual acuity testing as an objective measurement of macular oedema.

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant diabetic macular oedema involving the fovea in one or both eyes (phakic and/or pseudophakic) which persists at least 3 months after adequate macular photocoagulation.
* best corrected visual acuity in the affected eye(s) 6/9 or worse

Exclusion Criteria:

* Glaucoma which is uncontrolled or is controlled but with glaucomatous visual field defects
* Loss of vision due to other causes (e.g. age related macular degeneration, myopic macular degeneration)
* Significant macular ischemia (FFA)
* No useful vision in fellow eye
* Known allergies to triamcinolone acetate or steroids
* Patient is already under systemic treatment with > 5mg prednisolone (or equivalent) daily.
* Intercurrent severe disease such as septicaemia
* Any condition which would affect follow-up or photographic documentation (e.g. geographical, psycho-social, media opacities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2002-03; Study Completion 2005-04

PRIMARY OUTCOMES:
• Proportion of treated versus untreated eyes with improvement of visual acuity by 5 letters or more on the ETDRS chart at 24 months, no less than 3 months after the most recent treatment episode. An interim analysis of the primary and secondary outcome
• Incidence of moderate or severe adverse effects related to treatment

SECONDARY OUTCOMES:
• Any change of visual acuity (treated versus untreated eyes) at 3 months and 24 months after treatment
• Proportion of treated versus untreated eyes with reduction of macular thickness as demonstrated with OCT at 3 months and 24 months. Both absolute change and percentage change will be analysed.
• Changes in semi-quantitative grading of cataract at 3 months and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Gillies, MBBS, PhD, Principal Investigator — Save Sight Institute, Deaprtment of Clinical Ophthalmology, University of Sydney
Locations (1):
- Save Sight Institute, Sydney/Sydney Eye Hospital Campus, University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Result] Sutter FK, Simpson JM, Gillies MC. Intravitreal triamcinolone for diabetic macular edema that persists after laser treatment: three-month efficacy and safety results of a prospective, randomized, double-masked, placebo-controlled clinical trial. Ophthalmology. 2004 Nov;111(11):2044-9. doi: 10.1016/j.ophtha.2004.05.025. PMID 15522370
- [Result] Larsson J, Zhu M, Sutter F, Gillies MC. Relation between reduction of foveal thickness and visual acuity in diabetic macular edema treated with intravitreal triamcinolone. Am J Ophthalmol. 2005 May;139(5):802-6. doi: 10.1016/j.ajo.2004.12.054. PMID 15860283
- [Derived] Rittiphairoj T, Mir TA, Li T, Virgili G. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD005656. doi: 10.1002/14651858.CD005656.pub3. PMID 33206392
- [Derived] O'Day RF, Barthelmes D, Zhu M, Wong TY, McAllister IL, Arnold JJ, Gillies MC. Intraocular pressure rise is predictive of vision improvement after intravitreal triamcinolone acetonide for diabetic macular oedema: a retrospective analysis of data from a randomised controlled trial. BMC Ophthalmol. 2014 Oct 21;14:123. doi: 10.1186/1471-2415-14-123. PMID 25335434